CLINICAL TRIAL: NCT05247138
Title: Measurement of the Clinical and Radiological Performance Impact of the Root Canal Treatment With BioRootTM RCS: a Retro-prospective, National and Multicentre Clinical Study
Brief Title: Measurement of the Clinical and Radiological Performance Impact of the Root Canal Treatment With BioRootTM RCS.
Acronym: BioRoot
Status: Recruiting | Type: Observational
Sponsor: Septodont (Industry)
Collaborators: EndoData (Unknown); Recherche Clinique en Odontologie (ReCOL) (Network)
Responsible Party: Sponsor
Other Study IDs: BIOR 2021-04
Record Dates: First submitted 2021-12-28; First posted 2022-02-18 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Root Canal Obturation
Keywords: Root Canal Sealer; Endodontic Treatment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: BioRootTM RCS — BioRoot™ RCS is a hydrophilic mineral root canal sealer prepared from the mixture of a powder part and a liquid part. BioRoot™ RCS is a class III implantable medical device. This device is intended to be used in dentistry for permanent obturation of root canals of permanent and mature teeth with adjunction of gutta-percha points. Exposure to the sealer BioRootTM RCS starts from the day when the root canal treatment is performed until the end of individual observational period or the removal of the sealer in case of extraction or retreatment, if this event occurs before the end of individual observational period.

SUMMARY:
The aim of this retro-prospective Post-Market Clinical Follow-Up (PMCF) study is to collect long term clinical and safety data on root canal obturation after treatment, or retreatment, by BioRootTM RCS. The patients included in the study had received BioRootTM RCS 5 years ago. Participants will be followed prospectively at 5 and 10 years after root canal treatment.

Clinical data, radiographic data, adverse events (safety) and device performance will be collected by the dentist from the inclusion visit until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, > 18 years of age at the time of inclusion in the study.
* Patient who had a non-surgical root canal treatment with BioRootTM RCS, in a context of an endodontic treatment, or retreatment, 5 years (± 6 months) ago.
* All roots of the investigational teeth were treated with BioRootTM RCS.
* Having a documented retro-alveolar radiography immediately after root canal obturation.
* Patient affiliated or beneficiary of a social security system.
* Patient has signed his/her informed consent form.

Exclusion Criteria:

* History of malignant tumors in the 5 years prior to the root canal treatment.
* Non-stabilized systemic disease during the month prior to the root canal treatment (diabetes, hypertension, thyroid disorders, etc.).
* Patient who developed a systemic pathology after the root canal treatment with BioRootTM RCS.
* The Root canal treatment with BioRootTM RCS is on a wisdom tooth.
* Tooth presenting an advanced periodontal disease (parodontal pocket ≥ 5mm or bone loss ≥ 50%).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient in need of root canal treatment (or retreatment).
Sampling Method: Probability Sample
Enrollment: 142 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Clinical and radiological performance impact of the endodontic treatment at 5 years. | At 5 years post treatment
  The "success" and "failure" of the 5-year clinical and radiological performance impact of the endodontic treatment.

SECONDARY OUTCOMES:
Clinical and radiological performance impact of the endodontic treatment at 10 years. | At 10 years post treatment
  The "success" and "failure" of the 10-year clinical and radiological performance impact of the endodontic treatment.
  * Absence of pain
  * Absence of clinical evidence of infection, inflammation or swelling
  * Normal periodontal ligament space (PAI score ≤ 2)
    • "failure" of the endodontic treatment occur if the investigational tooth met one of the following criteria:
  * had been extracted for endodontic reasons since the root canal filling
  * Had been retreated since the root canal filling
  * Had undergone a periapical surgery since the root canal treatment
  * Presence of pain
  * Presence of clinical evidence of infection, inflammation or swelling
  * PAI score ≥ 3
Evaluation of the need of treatment or retreatment at 5 and 10 years. | At 5 and 10 Years post treatment
  "The "success" and "failure" of the endodontic treatment at 5 and 10 years according treatment or retreatment.
Assessment of the "tooth functional retention" at 5 and 10 years. | At 5 and 10 Years post treatment
  The success and failure of the "tooth functional retention" at 5 and 10 years after Root Canal Treatment with BioRoot™ RCS.
The technical characteristics of the sealer BioRootTM RCS at 5 and 10 years after Root Canal Treatment. | At 5 and 10 Years post treatment
  The technical characteristics of the sealer BioRootTM RCS at 5 and 10 years after Root Canal Treatment "Not resorbable once hardened", "Not retractable over the years" and "Radiopaque" will be evaluated in patients with retro-alveolar radiographs at the follow-up consultation (in parallel of the baseline consultation). The technical characteristics are defined as follows:
  * no resorption of the filling cement in the root, detectable on radiography
  * dense and homogeneous filling, limited to the canal
  * a filling with the maintenance of the canal anatomy
The ease of use and insertion of BioRootTM RCS in the canal. | At 5 years post treatment
  The ease of use and insertion of BioRootTM RCS in the canal will be evaluated with the score obtained on the Visual Analog Scale: score from 0 (Not at all) to 10 (Certainly Yes).
The Investigator overall satisfaction of the experience with BioRootTM RCS. | At 5 and 10 Years post treatment
  The Investigator overall satisfaction of the experience with BioRootTM RCS will be evaluated at 5 and 10 years after Root Canal Obturation with the score obtained on the Visual Analog Scale: score from 0 (Not at all) to 10 (Certainly Yes).
The post-obturation adverse device effects. | At baseline visit, 5 and 10 years post treatment
  The post-obturation adverse device effects will be evaluated with the list of adverse events occurring between the date of the root canal filling and the 5-year visit and between the 5-year visit and the 10-year visit.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Grosgogeat, MD, PhD, Study Director — CHU de Lyon, France
Locations (9):
- France (9):
  - Cabinet Dentaire, Levallois-Perret, Perret
  - Cabinet dentaire, Dijon
  - Cabinet Dentaire, Muizon
  - Cabinet dentaire, Muizon
  - Cabinet dentaire, Paris
  - Cabinet dentaire, Plérin
  - Cabinet dentaire, Saint-Amand-sur-Sèvre
  - Cabinet dentaire, Sézanne
  - Cabinet Medical, Villiers-sur-Marne

IPD SHARING:
Plan to Share IPD: No